CLINICAL TRIAL: NCT01552304
Title: The Benefit and Risk of Oxygen Supplementation in Perioperative Management of Obstructive Sleep Apnea
Brief Title: Oxygen Supplementation Study in Obstructive Sleep Apnea (OSA) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Dr. Frances Chung, Staff Anesthesiologist, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Protocol version May 30, 2011
Record Dates: First submitted 2012-03-06; First posted 2012-03-13 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2016-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea; Oxygen therapy; Surgery; Anesthesia
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Oxygen; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxygen treatment group (Experimental): Besides routine care, patients in this group will receive postoperative oxygen therapy with nasal prolong at 3 liters/min during the first 3 nights after surgery.
  Interventions: Other: Oxygen therapy
- Control group (Other): Patients will be managed by the anesthesiologists and surgeons as per routine practice.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Oxygen therapy — Besides perioperative routine care provided by anesthesiologists and surgeons, patients will receive postoperative oxygen supplementation with nasal prolong at 3 liters/min during the first 3 nights after surgery.
  Arms: Oxygen treatment group
Other: Control group
  Arms: Control group

SUMMARY:
Hypotheses:

1. Postoperative oxygen therapy significantly improves postoperative oxygenation in OSA surgical patients.
2. Postoperative oxygen therapy do not significantly increase the number of apnea episodes and the duration of apnea episodes.
3. Postoperative oxygen therapy do not significantly increase arterial carbon dioxide(CO2) level in OSA surgical patients.

DETAILED DESCRIPTION:
When patients visit the preoperative clinic for their scheduled surgery, the study coordinator will talk to patients. If they are interested in the study, he/she will ask the patient to answer a couple of questionnaires to see if the patient is qualified for the study. Patients will be asked to answer the STOP-Bang questionnaire to find out if patient is at high risk for sleep apnea. If the result shown that patient are at high risk for sleep apnea, the study coordinator will explain the study to you in detail and go over the consent form. The coordinator will answer all questions patient may have. If patient give consent to participate the study; the coordinator will schedule a sleep study with a sleep monitor at patient home at a convenient time before surgery. After telephone confirmation, the sleep technician will visit your home on the evening of scheduled date to set up the sleep study monitor and a device to measure the blood oxygen level. It would take 20~25 minutes to hook up for over night sleep study. The sleep technician will visit patient's again the next morning to pick up the devices. The recordings of sleep study will be scored by a certified sleep technologist. As a study participant, patient will be randomly (by chance) assigned into one of the following groups:

* Control group: Patients will be managed by the anesthesiologists and surgeons as per routine practice.
* Oxygen therapy group: Besides during surgical procedure routine care provided by anesthesiologists and surgeons, patients will receive postoperative oxygen supplementation with nasal prong (through nostril) at 3 liters/ min during the first 3 nights after surgery.

Regardless what group patients are in, their blood oxygen saturation will be monitored by a pulse oximeter for 1 night preoperatively and 3 nights postoperatively during their sleep. The blood carbon dioxide will be monitored for first 2 postoperative nights with a portable transcutaneous CO2 device (TCM400). On the third postoperative night, all study patients will also be monitored simultaneously by a portable carbon dioxide device(TCM400) and portable sleep device. For carbon dioxide monitoring, a probe will be attached to patient's arm which is connected to a portable device placed besides patient's bed. Our research staff will hook up the device and remove it from patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for inpatient surgery that requires a minimum of three nights of hospital stay
* Age: 18 to 80 years old.
* Identified as high risk of having OSA or diagnosed with OSA but not using CPAP.

Exclusion Criteria:

* Undergoing nasal, eye, head/neck surgery, intracranial or cardiac/thoracic surgery.
* Unwilling or unable to give informed consent.
* Requiring prolonged postoperative ventilation.
* Having chronic obstructive pulmonary disease,
* HCO3 ≥30.
* Visiting preoperative clinic < 1day before scheduled surgical date.
* Having tracheotomy, facial, neck, or chest wall abnormalities.
* Currently receiving treatment for sleep apnea including CPAP.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2012-02; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Pulse oxygen saturation | 3 nights postoperatively
  Nocturnal oxygen desaturation index and percentage of time with SaO2<90% on postoperative night 1 to 3.
Sleep disordered breathing | Postoperative night 3 only
  Including apnea hypopnea index, obstructive apnea index, central apnea index, hypopnea index, respiratory arousal index, and average and longest duration for obstructive, central and mixed apnea episodes, and hypopnea episodes on postoperative night 3.
Blood CO2 level | postoperative night1 to noght 3
  Transcutaneous CO2 level on postoperative night 1-3.

SECONDARY OUTCOMES:
perioperative clinical adverse events | 30 days after surgery
  Occurrence of perioperative clinical adverse events, especially cardiopulmonary adverse events.Intensive Care Unit(ICU) admission and ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Frances Chung, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Department of Aneshtesia, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Liao P, Wong J, Singh M, Wong DT, Islam S, Andrawes M, Shapiro CM, White DP, Chung F. Postoperative Oxygen Therapy in Patients With OSA: A Randomized Controlled Trial. Chest. 2017 Mar;151(3):597-611. doi: 10.1016/j.chest.2016.12.005. Epub 2016 Dec 19. PMID 28007620